CLINICAL TRIAL: NCT04812925
Title: A Phase 3, Multicenter, Open-Label, Long-Term Trial to Evaluate the Safety and Efficacy of Efgartigimod (ARGX-113) PH20 Subcutaneous in Adult Patients With Primary Immune Thrombocytopenia
Brief Title: A Phase 3 Study to Evaluate the Safety and Efficacy of Efgartigimod PH20 Subcutaneous in Adult Patients With Primary Immune Thrombocytopenia
Acronym: ADVANCE SC+
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2005
Record Dates: First submitted 2021-03-15; First posted 2021-03-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- efgartigimod PH20 SC (Experimental): Patients receiving efgartigimod PH20 SC treatment
  Interventions: Biological: efgartigimod PH20 SC

INTERVENTIONS:
Biological: efgartigimod PH20 SC — Subcutaneous injection with efgartigimod PH20 SC
  Other Names: ARGX-113 PH20 SC

SUMMARY:
A Phase 3 study to evaluate the safety and efficacy of efgartigimod PH20 subcutaneous in adult patients with primary immune thrombocytopenia

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the requirements of the trial and provide written informed consent (including consent for the use and disclosure of research-related health information), willing and able to comply with the trial protocol procedures (including attending the required trial visits).
2. Participants enrolled in the ARGX-113-2004 trial who completed the 24-week trial period.

Note: If a participant has had an SAE during the ARGX-113-2004 trial, their eligibility should be evaluated by the investigator and the sponsor's trial physician. The decision of enrolling the participant will be evaluated case by case.

3a. Agree to use contraceptives consistent with local regulations and the following:

• Female participants of childbearing potential must have a negative urine pregnancy test at baseline before receiving IMP.

In addition to the above criteria, for participants who want to continue receiving efgartigimod during an additional 52-week treatment period (only applicable in case efgartigimod is not yet commercially available for patients with primary ITP or available through another patient program for patients with primary ITP), the following criteria apply:

4. Ability to understand the requirements of the additional 52-week treatment period of the trial, to provide written informed consent (including consent for the use and disclosure of research-related health information), and to comply with the trial protocol procedures (including required trial visits).

5. Participant has completed a 52-week treatment period.

Exclusion criteria:

1. Introduction or continuation of nonpermitted medications during the ARGX-113-2004 trial (such as anti-CD20 therapy, romiplostim, monoclonal antibodies, Fc fusion proteins, or live/live-attenuated vaccines)
2. Use of any other investigational drug or participation in any other investigational trial
3. Known hypersensitivity reaction to efgartigimod PH20 SC or any of its excipients
4. Pregnant or lactating females and those who intend to become pregnant during the trial or within 90 days after last dose of efgartigimod PH20 SC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence, frequency, and severity of adverse events (AEs), AEs of special interest (AESIs), and serious AEs (SAEs) | 216 weeks
Vital sign measurement: blood pressure in the overall population | 216 weeks
ECG: PR, QT and QRS interval in the overall population | 216 weeks
Laboratory safety evaluations: CRP analysis in the overall population | 216 weeks

SECONDARY OUTCOMES:
Extent of disease control defined as the percentage of weeks in the trial with platelet counts of ≥50×10E9/L | 52 weeks
Proportion of patients with overall platelet count response defined as achieving a platelet count of ≥50×10E9/L on at least 4 occasions at any time during the 52-week treatment period | 52 weeks
Mean change from baseline in platelet count at each visit | 52 weeks
For patients rolling over from the ARGX-113-2004 trial with a platelet count of <30×10E9/L: time to response defined as the time to achieve 2 consecutive platelet counts of ≥50×10E9/L | 52 weeks
The percentage of weeks in the trial with platelet counts of ≥30×10E9/L and ≥20×10E9/L above baseline | 52 weeks
In patients with a baseline platelet count of <15×10E9/L in the current trial (ARGX-113-2005), the percentage of weeks in the trial with platelet counts of ≥30×10E9/L and ≥20×10E9/L above baseline | 52 weeks
In patients with the first exposure to efgartigimod PH20 SC, the proportion of patients who achieve a sustained platelet response defined as achieving platelet counts of ≥50×10E9/L for at least 4 of the 6 visits between week 19 and week 24 | 5 weeks (week 19-24)
In patients with the first exposure to efgartigimod PH20 SC, the proportion of patients achieving platelet counts of ≥50×10E9/L for at least 6 of the 8 visits between week 17 and week 24 | 7 weeks (week 17-24)
Proportion of patients for whom dose and/or frequency of concurrent ITP therapies have been reduced compared to baseline | 52 weeks
Rate of receipt of rescue therapy (rescue per patient per month) | 52 weeks
Incidence of the World Health Organization (WHO)-classified bleeding events | 52 weeks
Severity of the World Health Organization (WHO)-classified bleeding events | 52 weeks
Serum efgartigimod concentration observed predose (Ctrough) | 52 weeks
Change from baseline in PRO (Functional Assessment of Chronic Illness Therapy Fatigue Scale [FACIT-fatigue]) at planned visits | 52 weeks
Change from baseline in PRO (Functional Assessment of Cancer Therapy questionnaire-Th6 [FACT-Th6]) at planned visits | 52 weeks
Change from baseline in PRO (QoL (Short Form-36 [SF-36]) at planned visits | 52 weeks
Pharmacodynamics markers: total IgG | 52 weeks
Number of patients who performed self-administration at home over time | 52 weeks
Percentage of patients who performed self-administration at home over time | 52 weeks
Number of caregivers who administered the injection to the patient at home over time | 52 weeks
Percentage of caregivers who administered the injection to the patient at home over time | 52 weeks
Number of training visits needed for the participant or caregiver to be competent to start administering efgartigimod PH20 SC | 52 weeks
Number of self- or caregiver-supported administrations at home | 52 weeks
Percentage of self- or caregiver-supported administrations at home | 52 weeks
Incidence and prevalence of antibodies to efgartigimod | 216 weeks
Titers of antibodies to efgartigimod | 216 weeks
Presence of neutralizing antibodies (NAb) against efgartigimod | 216 weeks

CONTACTS AND LOCATIONS:
Locations (83):
- United States (5):
  - Investigator Site 0010116, Bentonville, Arkansas
  - Investigator site 0010045, Washington D.C., District of Columbia
  - Investigator Site 0010062, Fort Wayne, Indiana
  - Investigator site US0010042, Iowa City, Iowa
  - Investigator Site 0010095, Oklahoma City, Oklahoma
- Argentina (2):
  - Investigator Site 0540001, Buenos Aires
  - Investigator site 540004, Buenos Aires
- Australia (3):
  - Investigator Site 0610012, Garran
  - Investigator Site 0610003, West Perth
  - Investigator site 610005, Westmead
- Investigator Site 3590017, Plovdiv, Bulgaria
- Chile (3):
  - Investigator site 0560003, Reñaca
  - Investigator site 560002, Santiago
  - Investigator site 0560004, Temuco
- China (9):
  - Investigator site 860013, Beijing
  - Investigator Site 0860008, Bengbu
  - Investigator site 860055, Huizhou
  - Investigator Site 0860015, Shenzhen
  - Investigator Site 0860001, Tianjin
  - Investigator Site 0860010, Wuhan
  - Investigator Site 0860002, Wuxi
  - Investigator Site 0860011, Zhengzhou
  - Investigator site 860058, Zhenjiang
- Georgia (3):
  - Investigator Site 9950007, Tbilisi
  - Investigator site 9950009, Tbilisi
  - Investigator site 9950011, Tbilisi
- Greece (2):
  - Investigator site 300008, Athens
  - Investigator Site 0300009, Thessaloniki
- Investigator site 3530003, Dublin, Ireland
- Italy (4):
  - Investigator site 390043, Ferrara
  - Investigator Site 0390032, Milan
  - Investigator Site 0390044, Napoli
  - Investigator site 390041, Napoli
- Japan (7):
  - Investigator site JP0810015, Hirakata
  - Investigator Site 0810017, Iruma
  - Investigator Site 0810053, Kanagawa
  - Investigator Site 0810051, Kitakyushu
  - Investigator site 0810016, Shibukawa
  - Investigator site 810023, Shimotsuke
  - Investigator Site 0810038, Tama
- Investigator site 9620001, Irbid, Jordan
- Investigator site 520002, Aguascalientes, Mexico
- Investigator site 640005, Christchurch, New Zealand
- Investigator site 0470003, Sarpsborg, Norway
- Poland (3):
  - Investigator site PL0480013, Katowice
  - Investigator Site 0480026, Nowy Sącz
  - Investigator Site 0480037, Skorzewo
- Portugal (3):
  - Investigator Site 3510007, Lisbon
  - Investigator site 3510004, Porto
  - Investigator site 3510001, Vila Nova de Gaia
- Romania (3):
  - Investigator Site 0400005, Bucharest
  - Investigator site 400012, Bucharest
  - Investigator Site 0400007, Craiova
- Russia (4):
  - Investigator site 0070040, Kirov
  - Investigator Site 0070026, Moscow
  - Investigator Site 0070038, Nizhny Novgorod
  - Investigator Site 0070037, Novosibirsk
- South Africa (4):
  - Investigator site 270003, Johannesburg
  - Investigator site 270004, Observatory
  - Investigator site 270001, Pretoria
  - Investigator site 270002, Randburg
- South Korea (2):
  - Investigator site 820004, Seoul
  - Investigator site KO0820007, Seoul
- Thailand (6):
  - Investigator Site 0660002, Bangkok
  - Investigator Site 0660003, Bangkok
  - Investigator site 660005, Bangkok
  - Investigator Site 0660001, Bangkok Noi
  - Investigator site 0660004, Chiang Mai
  - Investigator site TH0660009, Khon Kaen
- Tunisia (2):
  - Investigator site 2610001, Sousse
  - Investigator site 2160002, Tunis
- Turkey (Türkiye) (9):
  - Investigator Site 0900007, Adapazarı
  - Investigator Site 0900003, Ankara
  - Investigator Site 0900008, Ankara
  - Investigator Site 0900015, Ankara
  - Investigator site 900004, Izmir
  - Investigator Site 0900014, Kocaeli
  - Investigator site 900010, Mersin
  - Investigator site 0900017, Tekirdağ
  - Investigator site 900019, Trabzon
- United Kingdom (3):
  - Investigator site 440005, Coventry
  - Investigator site UK044041, London
  - Investigator site UK0440014, Penzance

IPD SHARING:
Plan to Share IPD: Undecided